CLINICAL TRIAL: NCT00003820
Title: Phase 2 Trial to Evaluate the Efficacy of Anti-CD20 Antibody in Patients With Lymphocyte Predominant Hodgkin's Disease
Brief Title: Rituximab in Treating Patients With Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ranjana Advani (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ranjana Advani, Saul A. Rosenberg, MD, Professor of Lymphoma, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13452; 75967 (Other: Stanford IRB, historical); U2082N; LYMHD0003 (Other: OnCore)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma; Hodgkin Lymphoma (Category); Nodular Lymphocyte Predominant Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Rituximab; Biosimilar Pharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab 375 mg/m2 per week (Experimental): 375 mg/m2 rituximab by IV infusion weekly. The initial course of treatment is 4 weeks.
  Subjects who achieve an objective response or stable disease after the initial course (4 weeks) were permitted to continue additional 4-week cycles of treatment, for 3 additional courses starting every 6 months (ie, at 6; 12; and 18 months).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab (biosimilar is Zytux) is a chimeric monoclonal antibody against the protein CD20, which is primarily found on the surface of immune system B-cells. Rituximab destroys B-cells and is therefore used to treat diseases which are characterized by excessive numbers of B-cells, overactive B-cells, or dysfunctional B-cells. This includes many lymphomas, leukemias, transplant rejection, and autoimmune disorders.
  Other Names: Rituxan; MabThera; Anti-CD20; IDEC-C2B8; Zytux (biosimilar)

SUMMARY:
Phase 2 trial to study the effectiveness of rituximab in treating patients who have lymphocyte-predominant Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This study will evaluate the partial, complete, and overall response rates to rituximab of subjects with lymphocyte-predominant Hodgkin's lymphoma. Subjects will receive rituximab by IV infusion over several hours once a week for 4 weeks, followed by maintenance therapy as repeat course of the same dose and schedule rituximab at 6, 12, and 18 months.

This was a single-arm study with multiple treatment periods added by amendment (ie, Secondary Group), with results reported by treatment period. As this was always considered a single-arm study, there was no intent to report the results for the initial treatment period separately as the Initial Group vs the Secondary Group.

ELIGIBILITY:
INCLUSION CRITERIA

* Age ≥ 3 years
* Lymphocyte-predominant Hodgkin's disease (LPHD) of B-cell lineage
* Biopsy-confirmed expression of CD20 antigen
* At least one tumor mass measuring > 1.0 cm in largest dimension
* No evidence of active infection
* Subjects at high risk of Hepatitis B virus (HBV) infection should be screened prior to enrollment.
* Performance status of 0 to 2
* Absolute neutrophil count (ANC) > 1500/mL
* Platelet count > 50,000/mL
* Serum creatinine (Cr) < 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase < 2 x ULN, unless related to primary disease
* Bilirubin < 2 x ULN, unless related to primary disease
* Aspartate transaminase (AST) and alanine transaminase (ALT) < 2 x ULN, unless related to primary disease
* Subjects must be able to read and sign Institutional Review Board-approved informed consent

EXCLUSION CRITERIA

* Life expectancy at least 12 weeks
* Evidence of other active malignancies other than cured carcinomas in situ of the cervix or basal cell carcinoma of the skin
* Active HBV infection or hepatitis.
* Serious non-malignant disease (eg, congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections)
* Concomitant or treatment within prior 4 weeks with radiotherapy or chemotherapy (within prior 6 weeks for nitrosourea compounds)
* Concurrent treatment with prednisone or other systemic steroid medication
* Treatment with any investigational drug within 30 days prior to entry into the study
* Treatment with any investigational drug within 5 half-lives of that drug prior to entry into the study
* Major surgery, other than diagnostic surgery, within 4 weeks
* Any other conditions which, in the opinion of the investigator and/or sponsor, would compromise other protocol objectives
* Female patients must be of non-childbearing potential or using adequate contraception with a negative pregnancy test at study entry

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1999-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjana H Advani, MD, Study Director — Stanford University; Richard T Hoppe, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Advani RH, Horning SJ, Hoppe RT, Daadi S, Allen J, Natkunam Y, Bartlett NL. Mature results of a phase II study of rituximab therapy for nodular lymphocyte-predominant Hodgkin lymphoma. J Clin Oncol. 2014 Mar 20;32(9):912-8. doi: 10.1200/JCO.2013.53.2069. Epub 2014 Feb 10. PMID 24516013
- [Result] Horning SJ, Bartlett NL, Breslin S, et al. Results of a prospective phase II trial of limited and extended rituximab treatment in nodular lymphocyte predominant Hodgkin's disease (NLPHD). Blood [ASH Annual Meeting Abstracts]. 2007;110:abs644.

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 375 mg/m2 Per Week Inital Group: Rituximab 375 mg/m2 week by IV infusion for 4 consecutive weeks, every 6 months
  Initial Group of participants prior to the addition of the three extra cycle treatments.
- Rituximab 375 mg/m2 Per Week Secondary Group: Rituximab 375 mg/m2 week by IV infusion for 4 consecutive weeks, every 6 months
  Secondary Group of participants were added after the addition of the three extra cycle treatments.
Period: Cycle 1 (Initial Treatment)
Arm/Group | Rituximab 375 mg/m2 Per Week Inital Group | Rituximab 375 mg/m2 Per Week Secondary Group
Started | 23 | 16
Completed | 23 | 16
Not Completed | 0 | 0
Period: Cycle 2 (Maintenance Treatment)
Arm/Group | Rituximab 375 mg/m2 Per Week Inital Group | Rituximab 375 mg/m2 Per Week Secondary Group
Started | 0 (Initial Group of participants only received 1 cycle of treatment) | 16 (Pts with treatment response/stable disease at 6 mos, & eligible to continue.)
Completed | 0 | 16 (Patients with treatment assessment at 12 months)
Not Completed | 0 | 0
Period: Cycle 3 (Maintenance Treatment)
Arm/Group | Rituximab 375 mg/m2 Per Week Inital Group | Rituximab 375 mg/m2 Per Week Secondary Group
Started | 0 (Initial Group of participants only received 1 cycle of treatment) | 16 (Patients with treatment response/stable disease at 12 months)
Completed | 0 | 16 (Patients with treatment assessment at 18 months)
Not Completed | 0 | 0
Period: Cycle 4 (Maintenance Treatment)
Arm/Group | Rituximab 375 mg/m2 Per Week Inital Group | Rituximab 375 mg/m2 Per Week Secondary Group
Started | 0 (Initial Group of participants only received 1 cycle of treatment) | 16 (Patients with treatment response/stable disease at 18 months)
Completed | 0 | 16 (Patients with treatment assessment at 24 months)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a single-arm study with multiple treatment periods added by amendment (ie, Secondary Group), with results reported by treatment period. As this was always considered a single-arm study, there was no intent to report the results for the initial treatment period separately as the Initial Group vs the Secondary Group.
Groups:
- Rituximab 375 mg/m2 Per Week: Rituximab 375 mg/m2 per week by IV infusion for 4 consecutive weeks
Arm/Group | Rituximab 375 mg/m2 Per Week
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 37
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS, assessed as the number of patients 5 years after treatment who are alive and without a ≥ 50% increase from nadir in the sum of the product of the greatest lesion diameters (SPD) of any previously-identified abnormal node, or appearance of any new lesion
Time Frame: 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Rituximab 375 mg/m2 Per Week: Rituximab 375 mg/m2 week by IV infusion for 4 consecutive weeks every 6 months, for up to 4 treatment cycles
Arm/Group | Rituximab 375 mg/m2 Per Week
Number analyzed (Participants) | 39
participants | 18

2. Secondary Outcome: Overall Survival (OS)
Description: OS, assessed as the number of patients 5 years after treatment who are alive
Time Frame: 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Rituximab 375 mg/m2 Per Week: Rituximab 375 mg/m2 week by IV infusion for 4 consecutive weeks
Arm/Group | Rituximab 375 mg/m2 Per Week
Number analyzed (Participants) | 39
participants | 36

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response as assessed as Complete Response (CR) + Partial Response (PR)
  * CR was determined as complete metabolic response (CMR), meaning complete resolution of 18-fluorodeoxyglucose (FDG) uptake within the tumor volume so that it is indistinguishable from surrounding normal tissue.
  * PR was determined as partial metabolic response (PMR), meaning reduction of greater than 25% in the standardized uptake value (SUV) adjusted for body surface area (SUV-BSA). A reduction in the extent of tumor FDG uptake is not required for PMR.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- Rituximab 375 mg/m2 Per Week: 375 mg/m2 rituximab by IV infusion weekly, assessed after 4 weeks of treatment
Arm/Group | Rituximab 375 mg/m2 Per Week
Number analyzed (Participants) | 39
percentage of participants
  Overall Response (CR+PR) | 100
  Complete Response | 67
  Partial Response | 33

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Rituximab 375 mg/m2 Per Week: Rituximab 375 mg/m2 week by IV infusion for 4 consecutive weeks, every 6 months for 2 years.
  This was a single-arm study with multiple treatment periods added by amendment (ie, Secondary Group), with results reported by treatment period. As this was always considered a single-arm study, there was no intent to report the results for the initial treatment period separately as the Initial Group vs the Secondary Group.
Arm/Group | Rituximab 375 mg/m2 Per Week
Serious Adverse Events (participants affected / at risk) | 28/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab 375 mg/m2 Per Week (N=39)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer, metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Relapse/progressive disease, Hodgkin lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Relapse / transformation to aggressive B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab 375 mg/m2 Per Week (N=39)
Fatigue (General disorders) | 18 (19)
Pain (General disorders) | 20 (22) — Including: Abdominal, back, ear, knee, lower quadrant, hand, shoulder, thigh
Anemia (Blood and lymphatic system disorders) | 7 (7)
Abdominal bloating (Gastrointestinal disorders) | 1 (1)
Aches (General disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergy (Immune system disorders) | 8 (9)
Anxiety (Psychiatric disorders) | 4 (4)
Aphthous (Gastrointestinal disorders) | 1 (1)
Arm tingling (Nervous system disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Athlete's foot (Infections and infestations) | 1 (1)
Bloody stool (Gastrointestinal disorders) | 1 (1)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Buccal mucosa ulceration (Gastrointestinal disorders) | 1 (1)
Burning sensation (General disorders) | 1 (1) — from knee to feet
Cardiac disorder (Cardiac disorders) | 4 (4) — including: chest discomfort, chest heaviness, chest pain and chest tightness
Chills (General disorders) | 5 (5)
Claudication (Injury, poisoning and procedural complications) | 1 (1)
Cold (General disorders) | 2 (2) — Including: cold symptoms
Colon cancer (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Including: dry cough and/or with sputum
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Distress (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Double vision (Eye disorders) | 1 (1)
Dysesthesias (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Early satiety (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Elevated levels (Investigations) | 6 (6) — Including: cholesterol, glucose, Lactate dehydrogenase (LDH) and Prostate-Specific Antigen (PSA)
Epigastric gurgling (Gastrointestinal disorders) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1)
Facial hives (Immune system disorders) | 1 (1)
Feeling sleepy (Nervous system disorders) | 3 (3)
Fever (General disorders) | 7 (7)
Flushing (Immune system disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
GI bleeding (Gastrointestinal disorders) | 1 (1)
GI irritability (Gastrointestinal disorders) | 1 (1)
Graves hyperthyroidism (Endocrine disorders) | 1 (1)
Headaches (Nervous system disorders) | 6 (6)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Heart murmur (Cardiac disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hip bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 8 (8)
Indigestion (Metabolism and nutrition disorders) | 1 (1)
Infusion related reactions (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5)
Itching (Skin and subcutaneous tissue disorders) | 10 (10) — Including: Itchy ear, eye, face, nose , scalp and throat
arthralgias (Immune system disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Leukopenia (Investigations) | 1 (1)
Lymphopenia (Investigations) | 9 (9)
Maxillary sinus disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Memory loss (Nervous system disorders) | 1 (1)
Metastatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Morning stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgias (Immune system disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) — Including discharge
Nausea (Gastrointestinal disorders) | 4 (4)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Night sweats (General disorders) | 8 (8)
Numbness (Nervous system disorders) | 2 (2) — Including: numbness in hands and thighs
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral ulceration (Gastrointestinal disorders) | 1 (1)
Oropharyngeal ulceration (Gastrointestinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 2 (2)
Pressure in bilateral upper lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rhinitis (Infections and infestations) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right neck fullness (Endocrine disorders) | 1 (1)
Rigors (General disorders) | 4 (4)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scratchy throat (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Skin infection (Infections and infestations) | 2 (2) — Including: sores
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soreness in extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Superficial phlebitis (Vascular disorders) | 1 (1)
Swelling (Musculoskeletal and connective tissue disorders) | 4 (4)
Tightness in throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth abscess (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No